CLINICAL TRIAL: NCT06909214
Title: A Phase 4, Open-Label, Prospective, Single-Group, Multicenter Study to Evaluate the Clinical Outcomes of Efgartigimod PH20 SC in Adult Participants With New-Onset Generalized Myasthenia Gravis
Brief Title: A Study to Evaluate the Clinical Outcomes of Efgartigimod PH20 SC in Adults With New-onset Generalized Myasthenia Gravis (gMG)
Acronym: ADAPT-EARLY
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARGX-113-2407
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: New Onset Generalized Myasthenia Gravis (gMG)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Efgartigimod PH20 SC (Experimental): Participants receiving efgartigimod PH20 SC
  Interventions: Biological: Efgartigimod PH20 SC

INTERVENTIONS:
Biological: Efgartigimod PH20 SC — Subcutaneous injection of efgartigimod PH20 SC

SUMMARY:
The main purpose of this study is to measure how well adults with new-onset gMG (which means they've had generalized disease signs and/or symptoms for less than 1 year) respond to treatment with efgartigimod PH20 SC. The study consists of a treatment period of 51 weeks. The study duration for each participant will be approximately 58 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 18 years when signing the ICF
* Has been diagnosed with gMG of MGFA class II, III, or IV
* Is seropositive for AChR-Ab
* Is treatment-naive for gMG or has been administered AChEI for the treatment of gMG
* Had onset of generalized MG signs and/or symptoms within 12 months before screening; candidates who also had onset of ocular MG signs and/or symptoms within 24 months before screening may be enrolled in the study
* Has an MG-ADL score ≥5

Exclusion Criteria:

* gMG diagnosis of MGFA class I or V
* Underwent a thymectomy prior to screening, except thymectomy for treatment of nonmalignant thymoma prior to the gMG diagnosis
* Prior or current use of any of any systemic corticosteroid therapy or nonsteroidal immunosuppressive therapy for the treatment of gMG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-17 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who achieve MSE of MG at any time within the first 16 weeks of treatment with efgartigimod PH20 SC | up to 16 weeks
  MSE (minimal symptom expression) is defined as an MG-ADL (Myasthenia Gravis Activities of Daily Living) total score of 0 or 1. The MG-ADL scale assesses MG symptoms and their effects on daily activities. The score varies between 0 and 24 (with 24 the most severe).

SECONDARY OUTCOMES:
Changes from baseline in MG-ADL total scores over time | up to 51 weeks
  The MG-ADL (Myasthenia Gravis Activities of Daily Living) scale assesses MG symptoms and their effects on daily activities. The score varies between 0 and 24 (with 24 the most severe).
Changes from baseline in MG-QOL-15r total scores over time | up to 51 weeks
  The MG-QoL15r (Myasthenia Gravis Quality of Life 15-item scale revised) questionnaire is a patient-reported instrument that measures the impact of MG symptoms on Quality of Life. The score varies between 0 and 30 (with 30 the lowest quality of life).
Proportion of participants who are administered systemic corticosteroid therapy as background add-on therapy throughout the study | up to 55 weeks
Incidence of adverse events, serious adverse events and adverse events leading to study drug discontinuation | up to 55 weeks

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - University of California, San Diego - Altman Clinical and Translational Research Institute (ACTRI), La Jolla, California
  - Samir Macwan, M.D., Inc. (S corporation), Rancho Mirage, California
  - EZR Research, Boca Raton, Florida
  - University of Florida Jacksonville, Jacksonville, Florida
  - University of California Irvine, Orange, Florida
  - Medsol Clinical Research Center Inc, Port Charlotte, Florida
  - Baycare Medical Group, St. Petersburg, Florida
  - Emory Brain Health Center, Atlanta, Georgia
  - The Queen's Medical Center - West Oahu, Honolulu, Hawaii
  - Hawaii Pacific Neuroscience, Honolulu, Hawaii
  - HSHS Medical Group, O'Fallon, Illinois
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Visionary Investigators Network, Princeton, New Jersey
  - Cleveland Clinic, Cleveland, Ohio
  - Erlanger Neuroscience Institute, Chattanooga, Tennessee
  - Central Texas Neurology Consultants - Elligo, Round Rock, Texas

IPD SHARING:
Plan to Share IPD: No